CLINICAL TRIAL: NCT02214056
Title: Mobile Unit Screening of Pathologies Associated With Chronic Diseases - Part I Feasibility
Brief Title: Mobile Unit Screening of Pathologies Associated With Chronic Diseases - Feasibility
Acronym: DéProPAss
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/DC-02; 2013-A01703-42 (Other: RCB number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Type II Diabetes; Atherosclerosis
Keywords: mobile screening team; feasibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Patient Selection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: There is only one group in this study. Please see the inclusion/exclusion criteria.
  Intervention: Patient recruitment Intervention: Mobile team exam
  Interventions: Other: Patient recruitment; Procedure: Mobile team exam

INTERVENTIONS:
Other: Patient recruitment — Participating general practitioners (GPs) will inform and recruit participants from among regular patient consults. Using the provided web tools, GPs will organize a visit with the mobile team that fits the needs of the patient.
Procedure: Mobile team exam — Each patient enrolled will receive a standardized assessment in one locality, made in about two hours, and comprising:
  questionnaire responses, a complete physical exam, a 12-lead ECG, spirometry before and after administration of β2-agonists, an arterial Doppler ultrasound (carotid and abdominal), ankle-brachial index (systolic pressure at the toe).
  At the end of two hours, each patient will evaluate their satisfaction using a survey of acceptability and leave with a full report to the attention of their general practitioner (copy sent to Physician if needed) detailing the results of the different examinations.

SUMMARY:
The main objective of this study is to assess the feasibility of standardized screening for comorbidities among patients with one or more of three chronic diseases (diabetes, COPD, atherosclerosis) by a mobile unit at times and localities under-served by health actors.

DETAILED DESCRIPTION:
The investigators secondary objectives include assessing patient and GP satisfaction in relation to the mobile screening team.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has one or more of the following three diseases: (1) chronic obstructive pulmonary disease (COPD); (2) type II diabetes; (3) atherosclerosis.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* There is a need to take urgent therapeutic care in the opinion of the general practitioner
* The patient has received within the past year, a full examination including Doppler assessment of supra-aortic arteries, abdominal aorta and lower limbs; the patient has received a measure of the ankle-brachial index at the toe.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients at least 50 years of age with a chronic disease (COPD, Type II diabetes, atherosclerosis) recruited by one of the GP investigators.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible patients who actually received the mobile team exam | Day of mobile team exam (day 0)

SECONDARY OUTCOMES:
Observance: percentage of patients included that actually received the balance sheet | Day of mobile team exam (day 0)
Time in days between making the appointment by the general practitioner and the mobile team exam | Day of mobile team exam (day 0)
Average per patient time necessary to carry out the mobile team exam | Day of mobile team exam (day 0)
Average time required for the patient to fill out questionnaires | Day of mobile team exam (day 0)
Percentage of complete mobile team exams, that is to say in which all the data and all the variables have been collected and interpreted | Day of mobile team exam (day 0)
Percentage of GPs who participated in the study | Day of mobile team exam (day 0)
Percentage of mobile team exams in which one or more comorbidities was discovered | Day of mobile team exam (day 0)
GP and patient acceptability of the mobile team exam | Day of mobile team exam (day 0)
  Visual analog scales (ranging from 0 to 10) for access, delays, organization and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: David Costa, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (13):
- France (13):
  - Cabinet Médical - 47 rue de la République, Bessèges
  - Centre de Santé Médical, Bessèges
  - Centre médical des Olivettes, Ganges
  - Cabinet Médical - 5 rue Abbé Masson, La Grand-Combe
  - Cabinet Médical - 154 Place de la Poste, Lasalle
  - Cabinet Médical - Les Glycines, Lasalle
  - Cabinet Médical - Pont de Grammal, Molières-sur-Cèze
  - Cabinet Médical - 9 rue Racine, Nîmes
  - Cabinet Médical - 15 rue du Lac, Quissac
  - Cabinet Médical - 36 place de l'Esplanade, Saint-Ambroix
  - Centre Médical La Cantonnade, Saint-Florent-sur-Auzonnet
  - Cabinét Médical - 9 rue Villeneuve, Saint-Jean-du-Gard
  - Cabinet Médical - 7 bis avenue Rhin Danube, Sauve